CLINICAL TRIAL: NCT06572150
Title: Minimal Electrophysiology and Imaging Enhanced Deep Brain Stimulation (MIXT-DBS)
Brief Title: Minimal Electrophysiology and Imaging Enhanced Deep Brain Stimulation
Acronym: MIXT-DBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIXT-DBS
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Motor evoked potentials
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Intraoperative Electrophysiology (Experimental): Participants undergoing DBS for the diagnosis of Parkinson's disease
  Interventions: Procedure: Deep Brain Stimulation - Minimal Electrophysiology
- Standard Intraoperative Electrophysiology (Other): Participants who previously underwent DBS surgery for the diagnosis of Parkinson's disease
  Interventions: Procedure: Deep Brain Stimulation - Standard

INTERVENTIONS:
Procedure: Deep Brain Stimulation - Minimal Electrophysiology — Participants will undergo standard work-up and follow-up for DBS, but with minimal intraoperative electrophysiological testing.
  Arms: Minimal Intraoperative Electrophysiology
Procedure: Deep Brain Stimulation - Standard — Participants underwent DBS surgery with standard intraoperative electrophysiological testing.
  Arms: Standard Intraoperative Electrophysiology

SUMMARY:
The goal of this study is to learn if Deep Brain Stimulation (DBS) surgery can be streamlined for patients being treated for Parkinson's disease. The main questions it aims to answer are:

* Can a streamlined DBS surgery protocol with minimal electrophysiology and imaging (MiXT) safely replace the current use of intraoperative electrophysiology?
* Are we able to improve the efficiency, lower the invasiveness, and improve the clinical outcomes for patients undergoing DBS surgery?

Researchers will compare patients undergoing DBS surgery with this streamlined protocol to patients who previously underwent DBS surgery with the standard protocol to see if the accuracy, clinical outcomes, and efficiency improve.

Participants will undergo the standard protocol for DBS work-up and follow-up, but with minimal intraoperative electrophysiological testing.

DETAILED DESCRIPTION:
In deep brain stimulation (DBS), accurate implantation of the stimulation electrode into the surgical target is crucial for a successful clinical outcome. The classic technique for surgical planning uses stereotactic atlases developed from a limited number of post-mortem samples. To better account for individual variability, imaging- and electrophysiology-based techniques have been developed. Electrophysiological techniques may offer intraoperative insight into anatomical positioning. Macrostimulation and microelectrode recording are gold-standards for simulating the therapeutic effects of stimulation during surgery, as well as predicting the threshold of stimulation-induced side effects. However, these techniques result in increased procedural time, reduced accuracy due to brain shift, and increased procedural risk due to the up to five electrode penetrations through brain tissue for testing. Motor evoked potentials (MEPs) deliver stimulation across the test and final implanted electrode to predict distance to the motor tract, and have been previously shown by our group to be an effective predictor of therapeutic threshold and side effects.

High-resolution magnetic resonance imaging (MRI) may be used to directly visualize target structures for individual patients, such as the subthalamic nucleus (STN), internal globus pallidus (GPi), and ventral intermediate nucleus of the thalamus (VIM). However, differentiating between the target and surrounding tissue is challenging for some surgical targets, and pre-surgical MRI may give imprecise coordinates of brain structures due to brain shift during surgery. Advances in machine learning have led to the development of software for assisting with detecting surgical targets from MRI images and for merging intraoperative images with the preoperative MRI images to represent the stereotactic space and verify the electrode position within the operating room setting.

Currently, our center uses MEPs, microelectrode recordings, and macrostimulation with software and intraoperative imaging plan and conduct DBS surgeries. Macrostimulation and microelectrode recordings may be redundant with the introduction of intraoperative MEP testing. This study aims to assess the safety, accuracy and clinical outcomes of using the streamlined procedure of MEP testing with imaging and assistive software only. This technique will be referred to as the MiXT technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient qualifying for deep brain stimulation for the diagnosis of Parkinson's disease
* Informed consent

Exclusion Criteria:

* Lack of consent
* Electrical or other devices that preclude the performance of magnetic resonance imaging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of implanted electrode position | Intraoperative
  The distance between the final implanted electrode and the planned electrode, as measured on imaging software.

SECONDARY OUTCOMES:
Change in disease score units on the Unified Parkinson's Disease Rating Scale | Baseline, 12 months
  Assessment of therapeutic effects using the Unified Parkinson Disease Rating Scale
Change in disease score units on the Parkinsons Disease Questionnaire | Baseline, 12 months
  Assessment of therapeutic effects using the Parkinsons Disease Questionnaire
Efficiency of Surgery | Intraoperative
  Assessment of operating room times and length of stay in hospital
Intraoperative intensity of stimulation in milliampere | Intraoperative
  Intraoperative intensity of stimulation in milliamp, which elicits an activation of contralateral muscle groups (musculus interosseus dorsalis and the musculus tibialis anterior)
Safety of streamlined protocol | 4, 16, and 52 weeks post-surgery
  Number of adverse events (neurological deficits, infections, hemorrhages), hardware complications (e.g. electrode dislocation and breakage), psychiatric side effects (e.g. depression, hypomania, obsessive behaviour), and unexpected stimulation induced side effects

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Weise, MD, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth Health Science Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided